CLINICAL TRIAL: NCT01066091
Title: Postprandial Inflammatory Response in Healthy Men: Effect of Dietary Fat Source, Obesity and Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yves Boirie (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); ITERG (Industry)
Responsible Party: Sponsor-Investigator, Yves Boirie, MD, PhD, Pr Yves Boirie, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Organization: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: AU800; IDRCB 2009-A00322-55 (Registry Identifier: Afssaps); 05/2009 SWALRAND (Other: CRNH)
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2011-01

CONDITIONS: Healthy; Obesity
Keywords: Inflammatory response; High-fat meal; cytokines; Body composition
MeSH Terms: conditions — Obesity | interventions — Oleic Acid; Palmitic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- mashed potatoes (Placebo Comparator): Mashed potatoes is composed of potatoes and Skim milk powder.
  Interventions: Other: Mashed potatoes
- Mashed potatoes + Oleic Acid (Experimental): The test meal is mashed potatoes with 1g/Kg of weight of lipids with 75% of Oleic Acid
  Interventions: Other: Mashed potatoes + Oleic acid
- Mashed potatoes + Palmitic Acid (Experimental): The test meal is mashed potatoes with 1g/Kg of weight of lipids with 39% of saturated fat with 32% of palmitic acid.
  Interventions: Other: mashed potatoes + Palmitic acid

INTERVENTIONS:
Other: Mashed potatoes — Mashed potatoes: Potatoes + Skim milk powder
  Arms: mashed potatoes
Other: Mashed potatoes + Oleic acid — Mashed potatoes with 1g/Kg of weight, of lipids with 75% of Oleic Acid
  Arms: Mashed potatoes + Oleic Acid
Other: mashed potatoes + Palmitic acid — Mashed potatoes with 1g/Kg of weight, of lipids with 32% of palmitic acid
  Arms: Mashed potatoes + Palmitic Acid

SUMMARY:
The nature of dietary lipids, age and perivisceral adiposity could alter the postprandial inflammatory response. It is supposed that there is a relationship between the postprandial inflammatory response and the repartition of fat and lean mass, which could partially explain the muscle mass loss with age.

The aim of this study is to compare the inflammatory response of a normal meal or high fat meal (from different fatty acids sources) between young lean and young obese and aged lean and aged obese men.

DETAILED DESCRIPTION:
32 healthy volunteers will be separated into four groups: 8 young lean men, 8 young obese men, 8 aged lean men and 8 aged obese men. They will come to the center four times after inclusion, with 2 to 4 weeks wash out each time. At the first visit they will undergo different test to evaluate their body composition, glucose tolerance, resting energy expenditure, and muscular strength. At the other three visits, people will undergo a kinetic blood sampling, urine and biopsies of adipose tissue over a period of 8h after ingestion of a test meal. The different meals tested (Oleic acid vs palmitic acid vs no lipid) will be given in a random way over the three visits. Before each of these three visits, a controlled diet will be established. At the last visit body composition and muscular strength will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject giving his written informed consent
* Male from 20 to 35 years old and more than 60
* Affiliated to the French National Health Insurance
* Body mass index (BMI) ≤ 25kg/m² and waist circumference ≤94cm ; or BMI ≥ 28kg/m² and waist circumference ≥ 102cm.
* Complete blood count (CBC)-platelet, normal liver function and normal coagulation.
* Serology of Human immunodeficiency virus (HIV) and hepatitis C virus (HCV) negative
* normal Thyroid Stimulating Hormone(TSH)

Exclusion Criteria:

* Previous medical and/or surgery judged by the investigator as incompatible with this study
* Glaucoma
* C-reactive protein > 10 mg/l
* people over 120 kg
* People with triglyceridemia > 3 g/L or with familial hypercholesterolemia
* Fasting glycemia > 1,26 g/l, abnormal Oral Glucose Tolerance Test
* Dietary habits judged by the dietitian as incompatible with the study aim
* Vegetarians
* Nutritional allergies or xylocaïn allergy
* People with eating disorders
* Heavy consumer of alcohol or cigarette
* Practising intensive physical exercise
* People with medication that could interfere with the measured parameters: beta-blockers, statins, anticoagulants, antiplatelet agents, corticosteroids for more than 8 days.
* Depression or psychiatric treatment
* Being under someone's supervision
* Refusal to be registered on the National Volunteers Data file or refusal to sign the consent form
* Being in exclusion on the National Volunteers Data file
* Blood donation into the last two months preceding the study

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Inflammatory profile by interleukin-6 (IL6) concentration in plasma. | six times per day (kinetic: T0 to T480) on three interventional days

SECONDARY OUTCOMES:
Muscular strength, Body composition | Once at the first and at the last visit
Total plasma lipids (total cholesterol, HDL-Cholesterol, LDL-cholesterol, Triglycerides (TG), non-esterified fatty acid, Plasma hormonal profile, Plasma inflammatory profile, Markers of Endothelial function, Plasma lipopolysaccharide concentration. | Six times per day (kinetic: T0 to T480), on three interventional days
Pro-inflammatory cytokines expression in subcutaneous adipose tissue | Twice per day (before the meal and 6 hours after), on three interventional days
Urinary metabolomic profile | Three times per days (T0,T240,T480), on three interventional days

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, MD/PhD, Principal Investigator — CRNH; Stephane Walrand, PhD, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Human nutrition laboratory, Clermont-Ferrand, Auvergne, France

REFERENCES:
- See also: Related Info — http://www.inra.fr